CLINICAL TRIAL: NCT00832793
Title: Exploring the Learning Needs of Individuals With Inflammatory Arthritis From the Perspectives of Patients, Family Members and Friends, and Health Care Providers Patient Perspectives: Perspectives of Health Care Providers
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Mary J Bell, Sunnybrook Health Sciences Centre
Other Study IDs: DOCH2 449-2008
Record Dates: First submitted 2009-01-26; First posted 2009-01-30 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Arthritis
Keywords: Mixed methods research (qualitative and quantitative); Peer support; Early inflammatory arthritis; Self-management; Patient education
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Inflammatory arthritis (IA) is a major cause of long-term disability. Due to specialist shortages, failure of primary care providers and individuals to recognize the disease, and lack of awareness of the importance of early intervention, delays to rheumatologic care are common. Peer support models have been used for various health issues and may be one method to assist individuals with early IA to manage their disease and cope with stress. Qualitative research methods (one-on-one interviews) will seek out feedback on a peer support approach and explore the learning needs (informational needs, educational preferences) and opinions about emotional and appraisal support of individuals living with IA, from the perspectives of health care providers. The data will be analyzed and expressed themes (articulated needs and understandings of interviewee context) will guide the future development of a peer support intervention

DETAILED DESCRIPTION:
Abstract

Benefits of medical treatment in patients recently diagnosed with inflammatory arthritis are well documented, but delays in the commencement of these treatment regimens often leads to poor and irreversible healthcare outcomes. This study aims to explore the informational needs and educational preferences of persons with early inflammatory arthritis through the perspective of their health care providers in efforts to expedite the time to treatment. This project is part of a larger multidisciplinary study that also investigates these learning needs from the perspectives of the patients, their families, and their culture. Specifically for this part of the project, healthcare providers who are engaged in work related to inflammatory arthritis care will be invited to participate as key informants. Using a semi-structured interview guide, these participants will provide personal insight from their experiences in working with patients diagnosed with inflammatory arthritis regarding the informational and educational barriers they believe lead to delays in arthritis treatment in Ontario patients.

Rationale Disorders of the musculoskeletal system remain a prevalent cause of long-term disability in Canada and their burden on society and the health care system is projected to continue increasing1-5. There are currently over 4 million Canadians inflicted with arthritis, a figure projected to continue increasing to 6 million by 2026. Although there is currently no cure for this disease, medical intervention has been demonstrated to prevent disability, help maintain function, and reduce arthritis associated pain6.

Although the benefits of commencing early treatment in patients recently diagnosed with inflammatory arthritis are well documented6, delays due to the shortage in the number of qualified healthcare providers trained to meet the demands of this growing disease7-11 often leads to poor and irreversible health outcomes in these patients12-14. This disparity has created gaps in the care of these patients including access to arthritis-related services, specialist and rehabilitation services7,8. To compound this, the stress acquired following a diagnosis of inflammatory arthritis has been shown to greatly impede patients' cognitive function and decision-making abilities. Unlike the disparity in healthcare providers, these patient-related variables, although likely to play a major role in disease progression, are currently not well understood. In light of this, one cost-effective option to shortening the time between disease onset and treatment is to better understand the hurdles patients face following their diagnosis and develop more efficient mechanisms to deliver the information to this group more effectively. By exploring the informational needs and educational preferences of persons with early inflammatory arthritis, the development of such novel strategies will likely be possible.

Promoting patient education in self management encourages self-autonomy and is considered one of the key elements to optimal clinical practice. It increases confidence and self-esteem and empowers patients to be come more independent at coping and managing their arthritis15,16. Furthermore, self-management strategies increase the efficacy of prescribed medication and allow patients play a more active role in the management of their disease with relatively little supervision from healthcare providers17. These ideals are often not met in the clinical setting as a large proportion of patients fail to engage or continue with this independent approach. Such failures may be accounted for by the variable learning stages and individual needs of patients and thus require refinement in order to improve long-term adherence to self-management strategies18,19. Understanding the needs of patients in these different stages of learning will be vital to implement new patient-directed therapies.

Although, the wide array of different educational needs have yet to be systemically explored in a scientific manner, it is postulated one common problem in this patient population is a deterioration of sufficient self-confidence to make independent decisions. Onset of inflammatory arthritis leads to systemic profound fatigue, prolonged morning stiffness and severe joint pain compromising affected individuals' mood and ability to work and participate at home and in the community20. This alienation significantly decreases patients' independence and likely leads to subsequent increase in everyday stresses. Factors like these that greatly affect patient's learning and cognitive function need to be properly understood. One solution to this problem could involve the promotion of peer support in patients' lives and healthcare decisions20. Peer supporters are lay health advisers that offer encouragement and are seen as equal by the patients. The support often presents as one-on-one or focus groups between newly diagnosed patients and people who through personal or closely related encounters have previously been placed in similar decision making scenarios. They thus represent trusting figures that can easily sympathize with the difficult adjustments and decisions these patients need to make. Because of this connection, they often provide some degree of informational, appraisal and emotional support that other members of a healthcare team cannot. Such interventions that are designed to improve the social environment of individuals have been shown effectively improve psychological adjustment, recovery times and even extend the life expectancy of patients with chronic diseases20. Peer support is thus an important tool that when integrated into healthcare transforms the focus from disease treatment to overall health promotion21.

Understanding the education needs of the patients and their perceptions of peer support will likely lead to the development of better strategies that are more centered around patients. It is hoped that such novel strategies will play a key role in decreasing the diagnosis to treatment lag time currently affecting positive outcomes in the management of inflammatory arthritis.

The purpose of this study is to solicit the knowledge and experience of experts in the field (healthcare providers) working with inflammatory arthritis patients to develop a comprehensive understanding of strategies, including peer support that can be used to promote independence in the learning and decision making among patents with arthritis regarding their disease. Through dialog with these healthcare providers we hope to identify and better understand the barriers and facilitators in this process.

Purpose and Objectives The specific objectives of this phase of study are to explore the daily observations and personal experiences of different healthcare providers to identify the informational needs and educational preferences of persons with early inflammatory arthritis.

By conducting these interviews we hope to identify common hurdles and catalysts observed by healthcare providers preventing or promoting newly diagnosed inflammatory arthritis patients to make prompt decisions regarding the management of their disease. The aim is to identify processes important for the implementation and evaluation of the proposed model.

Methodology Through the perspectives of the healthcare providers, the informational needs and educational preferences for persons with early inflammatory arthritis will be explored using a qualitative approach. A sample size of approximately 10-15 health care providers (i.e. physicians, nurses, therapists) who are engaged in the management of inflammatory arthritis patients in Ontario will be asked to act as key informants. More specifically, this will be done through the use of both one-on-one in-person or telephone semi-structured interviews.

Study Design:

The semi-structured interviews will serve an as efficient investigation technique for assembling large amounts of data in a relatively short time frame that offers insight into a broad range of issues on a particular topic. A semi-structured interview guide (Appendix A) outlining the information that will be inquired about during the interview was developed for the purpose of this study. Semi-structured interviews entail asking each interviewee a specific set of predetermined questions in the same and consistent manner. However, they also allow flexibility for the interviewer to alter the order of the questions and probe the participants further to gain more information. These probes (or prompts) are questions not found in the interview guide that will be used to encourage elaboration of responses and further discussion to particular questions. These will be posed to the interviewees in a neutral and unbiased manner. Furthermore, additional questions may be added to subsequent interviews if deemed to be useful at extracting previously unanticipated and potentially useful information. Due to the qualitative nature of the study, the total number of participants is estimated to be between 10 and 15, and will depend on when saturation is achieved. Saturation occurs when no new information or emerging themes are uncovered with subsequent interviews. The interviews will be conducted by a medical student who is a co-investigator for the project and has undergone interview training from experienced researchers and are anticipated to last approximately one hour. During the interview, key points arising will be manually documented by the medical student. The completed interview will also be digitally audiotaped and transcribed verbatim, and the digital files, interview transcripts and field notes will be uploaded to a qualitative software package, NVivo 8.

Participants:

Potential study participants will be identified based on the following inclusion criteria:

1. Healthcare providers for patients diagnosed with inflammatory arthritis.
2. Physicians, nurses, occupational therapist, physiotherapists, social workers and other healthcare providers.
3. 18 years of age or older.
4. Able to participate in a 1 hour interview.
5. Ontario residents
6. Fluent in English

Recruitment and Consent Process:

The potential participants for this study will be identified as healthcare providers holding positions that offer experienced insight into the informational needs and educational preferences for patients recently diagnosed with early inflammatory arthritis. This may include physicians, nurses, physiotherapists, occupational therapists and social workers. These individuals will be selected based on inclusion criteria in through existing and emerging contacts with Dr. Mary Bell, a rheumatology physician at the Toronto General Hospital and Sunnybrook Health Sciences Centre. This initial contact will be made by Dr. Bell through e-mail, telephone, or personal contact. Recruitment will also take place through The Arthritis Society and using a snowball technique in which participants are asked to recommend others who could be contacted. An attempt will be made to select healthcare providers from different geographic locations (e.g. rural vs. urban) across Ontario.

Potential participants will be approached by the Principal Investigator (Dr. Mary Bell) and asked for their willingness to participate in this study. The individual will verbally agree to be contacted by the medical student who is a co-investigator with the project. Contact information of these potentially interested volunteers will be collected by the office manager at the clinic and then given to an experienced medical student responsible for obtaining consent and conducting the interviews. This medical student will obtain written consent and provide a copy to the participant. The medical student will then contact potential participants by telephone using a standardized telephone scripted (Appendix B) to further describe the study and re-confirm the willingness of the potential participants to take part in the study.

A confirmation letter (on Sunnybrook Health Sciences Centre letterhead, signed by Dr. Bell) with time and location of the interview/focus group will also be mailed to the participant (Appendix C). The day before the interview is scheduled to take place the medical student will telephone the individual to remind them of the time and location of the interview (Appendix D).

Interviews will be conducted by telephone or in person. The location and timing of the interviews will be conducted at a time and place that is convenient for each participant. If the participant lives or work in a remote rural area, if preferred, the interview will be conducted over the phone. Before each interview, participants will receive an information sheet describing the study (Appendix E) and a consent form (Appendix F) via e-mail, personal delivery or by mail. The information sheet will describe the purpose of the study, expected commitment for participation, the known benefits and risks of the study, and their right to refuse or withdraw at any time. The interview process will begin only after the participant has a chance to read over the forms and has an opportunity to ask questions about the study and consent process. Consent forms will be completed and signed by the participant prior to commencing the interview session. A photocopy of the form will be prepared for each participant for their records. If the interview is to be conducted over the phone, consent will be obtained from the participant in advance of the interview by fax or mail. With the interviewee's consent, the interview will be audio-recorded, and interviews will be transcribed in part or in whole for a more thorough analysis. Notes from the interview will be taken before, during and after the interview on an Interview Notes Form (Appendix G). In addition to notes on the interviewee's responses to the questions, comments will be made regarding the interviewer's personal thoughts on the interview itself, observations of any nonverbal communication, as well as conversations occurring before and after the interview itself (field notes). Audio files, interview transcripts and field notes will be uploaded to a qualitative software package, NVivo 8.

Data Analysis The data collected from the interviews will be analyzed using the constant comparative method and organized into themes. This process involves simplifying and categorizing the unique thoughts and descriptions given by the various interviewees' into common themes. This process will allow us to reduce and refer to the complexity of the information into more manageable and readily identifiable classes. These clusters aim to summarize what the significant and meaningful aspects of the data collected and allow for the proper interpretation and presentation of the data. The specific categories that will be used will be developed as an iterative process during the analysis of each interview and a coding scheme will be created. Categories will be added to the coding scheme until no further emerging themes can be identified. This analysis will be carried out by the medical student who conducted the interviews of the healthcare providers. To reduce any potential bias in the interpretation of the interviewees' responses, the interview transcripts will be independently coded by another person on the research team. Discussion between the two following the coding process will be used to reach a consensus on the emerging themes arising from each interview. The modifications made to the interview guide during the evolution of the study will be noted to ensure any discrepancies between information gathered from the initial participants and those near the end of the study.

Risks and Benefits There are no known risks associated with this study. In addition to possibly promoting awareness in healthcare providers participating in the study regarding their patient population, there may be indirect benefits to patients and providers due to the future care of individuals with inflammatory arthritis in Ontario. We will make the information freely available to allow other programs to also integrate the implications of our findings into their own practice.

Privacy and Confidentiality Only the principal investigator and research staff conducting the interviews will know the identity of the participants. No identifying information will be included on data collection forms. Upon agreement to partake in the study each participant will be assigned a unique study identification number. This ID number will be used to identify the occupation and responses of each participant. The list of names, addresses and phone number of each participant will be maintained in a password protected file at the department of rheumatology offices at Sunnybrook Health Sciences Centre. Only the principal investigator and research staff involved in the study will their associates will have access to this file. All information collected during the study will be strictly confidential. No names or identifying information will be used in subsequent publications or presentations. No identifying information will be shared with personnel not associated with the study or leave the confines of the hospitals involved in the study. Until their eventual destruction, all digital audio files and tangible copies of data will be stored in a locked research room at the Sunnybrook Health Sciences Centre. The data for this study will be retained for 25 years. A confidentiality agreement will be signed by the study coordinator and all second year medical students involved with the study.

Compensation Participants are recruited on a volunteer basis and there will be no monetary remuneration. The budget for this is outlined in Appendix H.

Communication of Results Dissemination of these results to study participants upon request (including interviewed healthcare providers) will be done through a working report. The findings in this report will also be communicated by the medical students to their peers and professors as a partial requirement for the completion of their "Determinants of Community Health" course. Upon completion, these results will also be shared to the public academic audience through publications and presentations of the findings.

Team Principal Investigator Dr. Mary Bell

Co-Investigator Joyce Nyhof Young Phedias Diamandis Romy Cho Lopa Das Chris Tran Paula Veinot

Study Coordinator Paula Veinot

Research Assistant Gaya Embuldeniya

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare providers for patients diagnosed with inflammatory arthritis.
2. Physicians, nurses, occupational therapist, physiotherapists, social workers and other healthcare providers.
3. 18 years of age or older.
4. Able to participate in a 1 hour interview.
5. Ontario residents
6. Fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health care providers of patients with inflammatory arthritis
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
learning needs (informational needs and educational preferences) | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] 1. Badley,E.M. J. Rheumatol. Suppl 43, 19-22 (1995). 2. Badley,E.M. & Wang,P.P. J. Rheumatol. 25, 138-144 (1998). 3. Badley,E.M., Rothman,L.M. & Wang,P.P. Arthritis Care Res. 11, 335-345 (1998). 4. Badley,E.M. & Wang,P.P. J. Rheumatol. 28, 1077-1082 (2001). 5. Perruccio,A.V., Power,J.D. & Badley,E.M. J. Rheumatol. 33, 1856-1862 (2006). 6. Schiff,M. Am. J. Med. 102, 11S-15S (1997). 7. Beaulieu,M., Choquette,D., Rahme,E., Bessette,L. & Carrier,R. Am. J. Manag. Care 10, 569-575 (2004). 8. Glazier,R.H. et al. J. Rheumatol. 30, 1846-1850 (2003). 9. Irvine,S., Munro,R. & Porter,D. Ann. Rheum. Dis. 58, 510-513 (1999). 10. Hernandez-Garcia,C. et al. J. Rheumatol. 27, 2323-2328 (2000). 11. Suter,L.G., Fraenkel,L. & Holmboe,E.S. Arthritis Rheum. 55, 300-305 (2006). 12. Anderson,J.J., Wells,G., Verhoeven,A.C. & Felson,D.T. Arthritis Rheum. 43, 22-29 (2000). 13. Wiles,N.J. et al. Arthritis Rheum. 44, 1033-1042 (2001). 14. Mottonen,T. et al. Arthritis Rheum. 46, 894-898 (2002). 15. Jordan,K.M. et al. Ann. Rheum. Dis. 62, 1145-1155 (2003). 16. Combe,B. et al. Ann. Rheum. Dis. 66, 34-45 (2007). 17. Keysor,J.J. et al. Critical review of arthritis self-management strategy use. Arthritis Rheum. 49, 724-731 (2003). 18. Kerns,R.D. & Habib,S. J. Pain 5, 357-367 (2004). 19. Keefe,F.J. et al. Pain 87, 303-313 (2000). 20. Dennis,C.L. Int. J. Nurs. Stud. 40, 321-332 (2003). 21. Cox,A.D. Br. J. Psychiatry 163, 6-18 (1993).